CLINICAL TRIAL: NCT04943952
Title: JZP458 -Asparaginase Erwinia Chrysanthemi (Recombinant) for the Treatment of Acute Lymphoblastic Leukemia (ALL) and Lymphoblastic Lymphoma (LBL) in Adult and Pediatric Patients Who Have Developed Hypersensitivity or Silent Inactivation to E. Coli-derived Asparaginase
Brief Title: JZP458 - Recombinant Erwinia Asparaginase for Treatment of ALL / LBL Patients With Hypersensitivity to E. Coli-derived Asparaginase
Status: Approved for marketing | Type: Expanded Access
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: JZP458-701-01
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma
Keywords: JZP458; Asparaginase Erwinia Chrysanthemi (Recombinant); Recombinant Erwinia Asparaginase; RC-P
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — asparaginase erwinia chrysanthemi recombinant

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Asparaginase Erwinia Chrysanthemi (recombinant) — Participants will receive JZP458 via intramuscular injection.
  Other Names: JZP458; RC-P

SUMMARY:
This study is an Expanded Access Protocol (EAP) of JZP458 in participants with ALL/LBL who are hypersensitive to an E.coli-derived asparaginase (allergic reaction or silent inactivation) and unable to access alternative licensed treatment, to receive JZP458 treatment prior to potential Food and Drug Administration (FDA) approval and commercial availability.

DETAILED DESCRIPTION:
JZP458 is a recombinant Erwinia asparaginase that utilizes a novel Pseudomonas fluorescent technology expression platform to produce an enzyme with no immunologic cross-reactivity to E.coli-derived asparaginases. JZP458 is currently being studied in an open-label, multicenter, dose confirmation, and Pharmacokinetic (PK) study of JZP458 in patients (of any age) with ALL/LBL who are hypersensitive to E. coli-derived asparaginases (allergic reaction or silent inactivation). This study is designed to assess tolerability and efficacy by measuring asparaginase activity. For the EAP, JZP458 will be provided free of charge by the Sponsor for the duration of the program. In addition, JZP458 will continue to be provided to eligible patients at referring sites until it becomes commercially available in the US.

JZP458 will be administered per each patient's original treatment plan, as long as the patient derives clinical benefit.

ELIGIBILITY:
Adult and pediatric patients with Acute Lymphoblastic Leukemia (ALL) or Lymphoblastic Lymphoma (LBL) who are hypersensitive to E.coli-derived asparaginases (allergic reaction or silent inactivation) and meet the criteria below:

Inclusion Criteria (Initial Requests):

* Patient (or parent/legally authorized representative thereof) is able to understand and voluntarily give informed consent/assent
* Patient has a diagnosis of ALL or LBL
* Patient received appropriate standard treatment without success (or no standard treatment exists for the patient's condition), and no satisfactory alternative drug is available
* Patient had a ≥ Grade 2 allergic reaction (Common Terminology Criteria for Adverse Events [CTCAE] v5.0) to a long-acting E. coli-derived asparaginase OR have silent inactivation
* Patient, in Investigators' opinion, has fully recovered from their prior allergic reaction to E. coli-derived asparaginase Note: Patients must have completed antihistamine, epinephrine, and/or corticosteroid treatment for the allergic reaction ≥ 24 hours prior to JZP458 administration.
* Patient has adequate liver function, defined as: direct (conjugated) bilirubin ≤ 3X upper limit of normal (ULN); serum glutamic pyruvic transaminase (SGPT)(alanine aminotransferase [ALT]), and serum glutamic-oxaloacetic transaminase (SGOT)(aspartate transaminase [AST]) ≤ 5X ULN
* For female patients of childbearing potential (i.e., fertile, following menarche) and male patients who have female partners of childbearing potential:

  * Patient has agreed to use medically acceptable methods of contraception with their partners for the duration of treatment with JZP458 and for 30 days after the last dose of JZP458.
  * Medically acceptable methods of contraception that the patient may use include abstinence, progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action; a combination of male condoms with either cap, diaphragm, or sponge with spermicide (double barrier methods).

Exclusion Criteria (Initial Requests):

* Patient is currently taking part in or is eligible for a clinical trial for JZP458
* Patient previously received asparaginase Erwinia Chrysanthemi AND has access to a short-acting non-E. Coliasparaginase
* Patient experienced concern of a possible adverse event (AE) related to asparaginase Erwinia Chrysanthemi
* Patient to receive asparaginase Erwinia Chrysanthemi within 1 week of plans to start JZP458
* Patient is concurrently receiving another investigational agent and/or treated with an investigational device at the same time as JZP458(within 48 hours)
* Patient has a history of ≥ Grade 3 pancreatitis (per CTCAE v5.0)
* Patient has a history of ≥ Grade 3 hypersensitivity to asparaginase Erwinia Chrysanthemi
* Patient has a prior history of asparaginase-associated ≥ Grade 3 (per CTCAE v5.0) haemorrhagic event or asparaginase-associated thrombus requiring anticoagulation therapy, excluding catheter-related thrombotic events
* Female patients who are lactating and do not agree to stop breast-feeding

Eligibility Criteria (Re-Supply Requests)

* Patient remains eligible for inclusion in the Expanded Access Protocol (EAP)
* Patient continues to benefit from treatment with JZP458
* Patient has not encountered unacceptable toxicity
* Patient has not shown signs/symptoms of relapsed or refractory disease
* Patient has not encountered ≥ Grade 3hypersensitivity symptoms
* Patient is not pregnant or breastfeeding

Sex: All
Age Groups: Child, Adult, Older Adult